CLINICAL TRIAL: NCT00766220
Title: Phase II Randomized Study of SIR-Spheres, Yttrium Microspheres With Cetuximab Plus Irinotecan for Patients With Advanced Colorectal Cancer Metastases to the Liver
Brief Title: Yttrium Microspheres With Cetuximab Plus Irinotecan for Patients With Advanced Colorectal Cancer Mets to Liver
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual and withdrawn/exclusion of 2 participants.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-0779
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Colon Cancer; Colorectal Cancer
Keywords: Colon; Liver; Colorectal cancer; Colorectal cancer metastases to the liver; Metastases to the liver; Colorectal cancer mets to liver; Colon cancer metastasized to liver; Yttrium microspheres; SIR-Spheres; Yttrium-90; Cetuximab; C225; Erbitux; IMC-C225; Irinotecan; CPT-11; Liver directed therapy
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Yttrium-90; Cetuximab; Irinotecan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SIR-Spheres + Therapy (Active Comparator): SIR-Spheres with Cetuximab + Irinotecan Therapy
  Interventions: Drug: SIR-spheres Agent Administration; Drug: Cetuximab; Drug: Irinotecan
- Therapy Only (Active Comparator): Cetuximab + Irinotecan Therapy
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: SIR-spheres Agent Administration — SIR-Spheres, resin microspheres containing pure Beta emitter Yttrium-90, given through femoral catheter over 10 minutes.
  Other Names: Yttrium-90; Yttrium 90; Yttrium microspheres
  Arms: SIR-Spheres + Therapy
Drug: Cetuximab — 400 mg/m2 by vein over 2 hours once a week.
  Cetuximab infusions will be continued weekly at a dose of 250 mg/m2 unless toxicity necessitates interruptions.
  Other Names: C225; Erbitux™; IMC-C225
Drug: Irinotecan — 350 mg/m2 (or 300 mg/m2 in patients who are greater or equal to 70 years of age, or have an ECOG PS of 2 or have had prior pelvic and/or abdominal irradiation), by vein over 90 minutes, every three weeks.
  Other Names: CPT-11

SUMMARY:
The goal of this clinical research study is to find out what effects radioactive particles, SIR-spheres, have when injected into the liver, followed by systemic chemotherapy with a combination of cetuximab and irinotecan compared to those who have systemic therapy alone, in patients with colon cancer that has metastasized to the liver. The safety of this treatment and how well it controls the disease will also be studied.

DETAILED DESCRIPTION:
Yttrium microspheres are designed to treat cancer that has metastasized to the liver by giving radiation directly to the tumor. SIR-spheres are designed to deliver radiation directly to the tumor. This radiation kills the tumor cells.

Cetuximab is a drug that blocks epidermal growth factor receptor (EGFR). EGFR may be involved in certain types of cancer, including non small-cell lung cancer (NSCLC). When EGFR is stimulated, a series of chemical reactions start that result in a tumor being "told" to grow. Cetuximab tries to stop these reactions by blocking EGFR. This may stop tumors from growing.

Irinotecan is designed to block cell growth by blocking an enzyme that repairs DNA, the building blocks of cells.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1of 2 groups. Participants in one group will receive the SIR-spheres with Cetuximab and Irinotecan therapy. Participants in the other group will just have the Cetuximab and Irinotecan therapy without the SIR-spheres. There is an equal chance of being assigned to either group.

If you are found to be eligible to take part in this study, you will have a blood vessel study (given with x-ray dye) performed. This will help researchers look at the arteries leading to your liver and the surrounding areas. You will receive Versed and Fentanyl, sedative drugs to put you to sleep, intravenously (IV--through a needle in a vein) in your arm. A catheter will be placed through your groin artery into the artery leading to your liver. A catheter is a sterile flexible tube that will be placed into a large artery while you are under local anesthesia and IV sedation. Your physician will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure. X-ray dye will be injected through the catheter.

If randomly selected to receive the SIR-Spheres with Cetuximab and Irinotecan therapy, a small amount of radioactive albumin injection (a part of a scan test used to measure the supply of blood through the lungs) will be given to your liver. Images will then be taken to learn if too much of this material (radioactive particles) shows up in your lungs and if your liver anatomy is normal. If everything appears normal, the yttrium microspheres will be given slowly through the catheter in 1 dose. If your liver anatomy is abnormal, the yttrium microspheres will be given slowly through the catheter in 2 doses. After you are given the yttrium microspheres, the catheter will be removed, and pressure will be applied to your groin to stop any bleeding. You will then be monitored for 6 hours to check on your well being. You will be given pain medication, if needed (the same sedative drugs used before).

You will be given standard doses of Zantac (ranitidine) to help to protect the stomach during treatment. Chemotherapy with cetuximab and irinotecan will be given on an outpatient basis. A catheter (PICC line, port-a-cath) may be inserted through a vein in your arm or chest to ensure that the chemotherapy is given without interruption. Irinotecan will be given by IV over 90 minutes, once every 3 weeks. Cetuximab will be given once a week. On Day 1 of treatment, you will be given a test dose of cetuximab, to check for any allergic reactions. After that, cetuximab will be given by IV over 2 hours. Before every dose of cetuximab, you will be given a dose of diphenhydramine by IV, to keep from having any allergic reactions. You will also receive medication to prevent nausea, vomiting, or an allergic reaction.

You will have a single-photon emission computerized tomography (SPECT) scan within 1 week after your treatment. A SPECT scan lets your doctor study the function of your internal organs. You will have blood (about 2 tablespoons) drawn every week for the first 2 months and then once a month on an outpatient basis. This is so researchers can check the function of your kidneys and liver. You will also have a routine physical exam and a computerized tomography (CT) scan performed once a month to check the growth of your tumor. Researchers will check to see if your tumor is responding to the study treatment by looking at the imaging on CT scans every 8 weeks.

You may be taken off this study if your disease gets worse, if you experience intolerable side effects, or if there is not enough of the study drug supply to continue treating your disease.

You will be followed-up by telephone for as long as you have cancer.

This is an investigational study. Yttrium microspheres are FDA approved for hepatic arterial therapy and treatment of liver metastases. Sir-Sphere therapy has been approved for treating colorectal cancer with liver metastases. The combination of cetuximab and irinotecan is FDA approved for metastatic colorectal cancer. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the colon or rectum. Histology from the hepatic metastasis is not mandatory if the morphological appearances on cross sectional imaging and tumor markers (CEA) are indicative of a colorectal primary.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in two dimensions (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT scan.
3. Patients must have radiological evidence of disease progression of disease within 6 months of their most recent dose of chemotherapeutic regimens .
4. Age greater than or equal to 18 years.
5. ECOG performance status less than or equal to 2.
6. Patients must have normal organ and marrow function as defined below within 30 days of receiving the investigational agent: - leukocytes greater than or equal to 3,000/mL - absolute neutrophil count greater than or equal to 1,500/mL - platelets greater than or equal to 100,000/mL - total bilirubin less than or equal to 1.5 times upper limits of normal institutional limits - AST(SGOT) less than or equal to 3 X ULN and ALT(SGPT) less than or equal to 3 X ULN - Creatinine less than or equal to 1.5 times upper limits of normal institutional limits
7. Patients with a prior history of non-colorectal cancer who have no active disease may be eligible if they are disease free for greater than or equal to 12 months prior to treatment.
8. The effects of SIR-Spheres, irinotecan or cetuximab on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because radiation as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.
9. Ability to understand and the willingness to sign a written informed consent document.
10. Patients without evidence of local disease recurrence from colorectal cancer are eligible
11. Patients with extrahepatic disease confined to the lung is permitted if < 4 lesions are depicted on CTand all are < 3 cm in size
12. Patients with brain mets are eligible for this trial if those patients who have had the area surgically resected or irradiated and have no evidence of active disease as demonstrated by MRI of the brain. Patients must have no evidence of residual neurological dysfunction as per baseline neurological exam. Patients with untreated brain metastases will be considered ineligible.

Exclusion Criteria:

1. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier will be excluded. Patients who have had hepatic external beam radiotherapy will be excluded.
2. Patients may not be receiving any other investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to SIR-Spheres, irinotecan or cetuximab or other agents used in the study.
4. Evidence of ascites, biopsy proven cirrhosis or portal hypertension suggested by the presence of characteristic imaging features on cross sectional imaging or esophageal varicosities demonstrated on endoscopy or barium swallow. A diagnostic study to rule out the presence of portal hypertension will not be required unless the findings on cross sectional imaging are suggestive but not confirmatory.
5. Hepatic arterial anatomy that would prevent catheterization and the administration of SIR-Spheres into the liver.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring hospital admission or antibiotics,symptomatic congestive heart failure (class III and IV), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations would exclude patients from this study.
7. Contraindications to angiography and selective visceral catheterization: History of severe allergy or intolerance to any contrast media, or atropine. Bleeding diathesis, not correctable by usual forms of therapy that would include medical coagulopathy but not limited to the administration of blood products.
8. Utilization of capecitabine for the 6 weeks preceding SIR-Sphere therapy and indefinitely following SIR-Sphere therapy as per manufacturer's recommendations due to the increased risk of radiation hepatitis.
9. Patients exhibiting the mutant variety for kras will be excluded for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Murthy, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org